CLINICAL TRIAL: NCT06001320
Title: Historical Controlled, Single Center Open Label Pilot Comparing the Effectiveness and Tolerability of De-novo Initiation of Letermovir Versus Valganciclovir for Cytomegalovirus Prophylaxis in AA Kidney Transplant Recipients
Brief Title: De-novo Initiation of Letermovir vs Valganciclovir for Cytomegalovirus Prophylaxis in AA Kidney Transplant Recipients
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HM20027540
Record Dates: First submitted 2023-07-18; First posted 2023-08-21 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Kidney Transplant; Complications; CMV
MeSH Terms: interventions — letermovir; Health Records, Personal

STUDY DESIGN:
Intervention Model Description: Interventional, Historical Controlled, Single Center Open Label Pilot Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Letermovir group (study group) (Experimental): Letermovir 480 mg once daily
  Interventions: Drug: Letermovir 480 mg once daily
- Historical Control study group (Other): Historically matched AA kidney transplant recipients who received the standard of care 450mg once a day valganciclovir prophylaxis
  Interventions: Other: Historical/Control

INTERVENTIONS:
Drug: Letermovir 480 mg once daily — We will test the study hypothesis in a single center, matched (1:1 fashion) pilot study of Letermovir 480 mg once daily versus historically matched AA kidney transplant recipients who received valganciclovir. We will enroll 30 AA patients over a 12-month period into the Letermovir group and compare outcomes to a historical group of 30 AA kidney transplant recipients who have received valganciclovir prophylaxis (1:1 fashion), for a total of 60 patients. We will attempt to match patients on Letermovir to the historical patients who received valganciclovir, based on age, kidney Donor profile index and the presence of panel of reactive antibodies.
  Arms: Letermovir group (study group)
Other: Historical/Control — The control study group will include high-risk African American kidney transplant recipients cared for with Valganciclovir in the 5 years prior to the enrollment start for the study group. This time frame is based upon the current volume of transplants done at VCU. On average 30 liver and/or kidney transplants are done per month. Thus, 5 years should be an adequate time frame to mine enough number of participants to answer our primary research hypothesis.
  Arms: Historical Control study group

SUMMARY:
This study is being done to compare the effectiveness of de novo Letermovir versus valganciclovir in preventing the development of cytomegalovirus viremia or symptomatic disease in African American kidney transplant recipients within the first year after transplantation.

There are two arms in the study:

Arm 1: Prophylaxis: This group includes freshly transplanted high risk (CMV D+/R-) African American Kidney recipients who will be on prophylactic Letermovir for 6 month.

Arm 2: Prophylaxis: This group includes high-risk African American kidney transplant recipients who had already completed the 6 month prophylactic course with the standard of care Valganciclovir.

DETAILED DESCRIPTION:
Valganciclovir (VGC) is the drug of choice for CMV prophylaxis. Although effective in preventing CMV infections, VGC is commonly associated with profound bone marrow suppression, specifically leukopenia which increases patients' vulnerability to other infections. Moreover, kidney transplant recipients often receive lymphocytic antibody therapy for induction immunosuppression, which further exacerbates the risk of leukopenia in the first 3-6 months after transplantation. The high leukopenia burden makes management of immunosuppression in the post-transplant setting more complex, often necessitating reduction in immunosuppressive agents that increases risk of allograft rejection.

Primary Objective: this study is being done to compare the effectiveness of de novo Letermovir versus the standard of care valganciclovir in preventing the development of cytomegalovirus viremia (defined as CMV PCR > 137 units/ml) or symptomatic disease in AA kidney transplant recipients within the first year after transplantation.

Secondary Objectives: included leukopenia incidence, acute rejection rates, breakthrough CMV rates, mycophenolate dose adjustments, donor-specific antibody formation, and tolerability.

To compare these these two groups the study uses

* Intervention Letermovir: Recipients in this group will be on prophylactic Letermovir 480mg once a day pill started within the first 5 days of post-transplant up until 6 months post-transplant. Given Letermovir has no activity against herpes viruses, solid organ transplant recipients are at risk of herpes simplex viruses. Participants enrolled in this study group will also receive prophylactic acyclovir 400mg twice daily for the duration of their Letermovir treatment. Both Letermovir and study mandated medication (Acyclovir) are already approved for use by the FDA.
* Intervention Valganciclovir- In this group recipients who have historically received the standard of care prophylactic valganciclovir will be assessed retrospectively. Valganciclovir is 450mg once a day pill started with in the first 10 days post-transplant or at the time of discharge after kidney transplant and taken up until 6 month post-transplant. This historical control study group will include high-risk African American kidney transplant recipients identified from prior research studies who were cared for with Valganciclovir in the 5 years prior to the enrollment start for the study group.

Outcomes of these two groups will be compared in 1:1 fashion. The study will attempt to match patients on Letermovir to the historical patients who received valganciclovir, based on age, kidney Donor profile index and the presence of panel of reactive antibodies.

Strategy for CMV Viremia: CMV viremia will be treated with either oral valganciclovir, intravenous ganciclovir or alternative agents, according to AST ID COP (American Society of Transplantation Infectious disease community of practice) guidelines.

ELIGIBILITY:
Historical Control group:

Inclusion Criteria

1. Kidney transplant recipients
2. Male or female age ≥ 18 years old
3. African American race
4. CMV high risk (D+/R-)
5. received valganciclovir for CMV prophylaxis

Historical Control group:

Exclusion

1. Re-transplantation
2. Panel of reactive antibody ≥80% at the time of transplant
3. Positive cytotoxic cross match at the time of transplant

Experimental Group Inclusion Criteria

1. Kidney transplant recipients
2. Male or female age ≥ 18 years old
3. African American race
4. CMV high risk (D+/R-)
5. Ability to provide informed consent before any trial related activities

Exclusion Criteria

1. Re-transplantation
2. Panel of reactive antibody ≥80% at the time of transplant
3. Positive cytotoxic cross match at the time of transplant
4. Pregnancy and Breastfeeding
5. Prisoners
6. Patients with hypersensitivity to acyclovir, valacyclovir or any of its components
7. Patients with hypersensitivity to Letermovir or any of its components
8. If Patients are taking any of these medications: pimozide, ergot alkaloids (ergotamine, dihydroergotamine), or pitavastatin/simvastatin co-administered with cyclosporine, we will work with the prescribing physician to find an appropriate replacement therapy which will not interfere with any study-related interventions. Otherwise, participants will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of cytomegalovirus viremia (defined as CMV PCR > 137 units/ml) or symptomatic disease in AA kidney transplant recipients | up to one year after transplantation
  The incidence of cytomegalovirus viremia (defined as CMV PCR > 137 units/ml) or symptomatic disease in AA kidney transplant recipients by one year post-transplantation

SECONDARY OUTCOMES:
Incidence of Leukopenia (defined as WBC < 2.5 x 103 cells/mm3 beyond the first 2 weeks of transplantation, while on pharmacologic CMV prophylaxis) | From 2 weeks up to 26 weeks post-transplant
  The incidence of leukopenia (defined as WBC < 2.5 x 103 cells/mm3 beyond the first 2 weeks of transplantation, while on pharmacologic CMV prophylaxis)- assessed from 2 weeks up to 26weeks post-transplant
Impact of Pharmacological Prophylaxis on CMV T-Cell immunity up to 1 year post-transplant | up to 1 Year post-transplant
  CMV T-cell immunity assay, assessed up to 1 year post-transplant. At 12, 26 and 52 weeks post-transplant
Incidence of acute kidney allograft rejection up to one year after transplantation | up to 1 Year post-transplant
  acute kidney allograft rejection up to one year after transplantation
Impact of Pharmacologic CMV Prophylaxis on Mycophenolate dosage up to 6 months post-transplant | Up to 6 months post-transplant
  Changes in mycophenolate dosage (assessed by review of patient's chart) up to 6 months post-transplant
Incidence of de novo donor specific antibody formation up to 1 year after transplant | up to 1 Year post-transplant
  de novo donor specific antibody formation up to one year after transplantation
Tolerability of Letermovir in AA kidney transplant recipients up to 6 months post-transplant using a tolerability assessment questionnaire | up to 6 months post-transplant
  Tolerability of Letermovir in AA kidney transplant recipient up to 6 months post-transplant (assessed through patient observation, tolerability assessment questionnaire, obtaining medical history and conduction physical examination during visits, receiving an unsolicited complaint from the participant, and an abnormal value or result from a clinical or laboratory evaluation).
Correlation between CYP3A5*1 and its impact on tacrolimus metabolism and incidence of kidney allograft rejection up to 1 year post-transplant | up to 1 Year post-transplant
  correlation between CYP3A5*1 and tacrolimus metabolism and incidence of kidney allograft rejection up to one year after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav Gupta, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- VCU Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No